CLINICAL TRIAL: NCT03185754
Title: Comparison of Sublobar Resection and Lobectomy to Treat Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201212107RIND
Record Dates: First submitted 2013-06-13; First posted 2017-06-14 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Lung Cancer; Surgery
Keywords: lung cancer; surgery; lobectomy; sublobar resection
MeSH Terms: conditions — Lung Neoplasms | interventions — Anterior Temporal Lobectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- early phase lung cancer (Experimental): sublobar resection and lobectomy
  Interventions: Procedure: Sublobar resection; Procedure: lobectomy

INTERVENTIONS:
Procedure: Sublobar resection — Sublobar resection
Procedure: lobectomy — lobectomy

SUMMARY:
A multi-center prospective randomized trial in Taiwan to investigate whether sublobar resection, as compared to lobectomy, can offer equivalent clinical results to treat early non-small cell lung cancer.

DETAILED DESCRIPTION:
Background: Lung cancer has become an important disease threatening the public health world-wide. Surgical resection is the standard of care for treating non-small cell lung cancer in early stage. For decades, pulmonary lobectomy with lymph node dissection remains the gold standard of surgical approach. Pulmonary sublobar resection with pulmonary wedge resection or segmentectomy was reserved for the patients with high surgical risk, who were unsuitable for radical surgical resection. Pulmonary sublobar resection for tumor less than three centimeter was demonstrated to associated with higher risk of tumor recurrence or worsening survival outcome as compared to that done by lobectomy. 1 However, these data was which was not necessarily applicable to patients with early lung cancer with tumor of smaller size which was more frequently detected with the health screening test by CT scan in general population now. Although several retrospective studies has demonstrated that sublobar resection can offer a similar survival outcome after surgery as compared to that done by standard lobectomy once the tumor was smaller than two centimeter 2, there is still no consensus about the role of sublobar resection for these small early lung cancer. In general, there are several factors associating with higher risk of local recurrence which should be avoided for sublobar resection, including resection margin less than 2 cm or less than the diameter of the tumor itself 3, more obvious speculation in CT image or central location which makes it difficult to obtain adequate resection margin 4,5. Therefore, sublobar resection should be applied to the patients of early lung cancer when two cm of resection margin is achievable. The central location , obvious tumor infiltration in image study or presence of lymph node metastasis should be also avoided.

Patients and methods: The study will include surgical patients from six medical centers in Taiwan. All of the patients will receive complete study about the surgical risk and tumor staging before surgery. The patients will receive general anesthesia and pulmonary resection as the standard procedures including division of pulmonary vessels and bronchus. Either VATS (Video-assisted thoracoscopic surgery) or open surgery is acceptable for the surgical approaches. The patients will be randomly assigned to lobectomy and sublobar resection groups. Two cm of resection margin will be obtained in each patient in the sublobar resection group by wedge resection or segmentectomy. Standard lymph node dissection including the pulmonary hilum and mediastinum will be done in both groups of patients. For suspicious of pulmonary hilum or mediastinal lymph node metastasis, frozen pathological examination will be requested.

Post operative care and follow-up: The patients will be transferred to intensive care unit or surgical recovery room after surgery. Medication for pain control and postoperative rehabilitation education will be given to each patient after surgery. The chest tube will be removed after daily discharge less than 100 to 200 ml without air-leakage, adequate lung expansion noted in chest X ray imaging. The patient will be discharged from the hospital one or two days after removal of the chest tube. Whole body bone scan and CT scan will be given in every 6 months at least after surgery for postoperative follow-up.

ELIGIBILITY:
Inclusion criteria:

* Early non-small cell lung cancer (stage Ia) with diameter of two centimeters or less.
* Tumor locating at the peripheral lung parenchyma (outer one third in CT imaging).
* No suspected hilar or mediastinal lymph nodes metastasis in the CT or PET imaging study.

Exclusion criteria:

* Tumor diameter more than 2 centimeter
* Hilar or mediastinal lymphnode metastasis by the cancer.
* Patients received previous surgery in the ipsi-lateral lung
* Lung tumor locating in the central lung parenchyma unable to obtain curative resection by sublobar resection.
* Patients with poor cardiopulmonary function unsuitable for receiving surgical resection.
* Patients who have multiple lung cancer or other suspicious lesion in the lung.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-06-12 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 5 years
  The time interval from randomization to the earliest onset of any of the following events: tumor local recurrence, distant metastasis, and mortality

SECONDARY OUTCOMES:
post-operative complication | 3 months
  defined as any deviation from the normal postoperative course
Hospitalization time | 3 months
  the time interval from the day of surgery to discharge
Chest tube duration | 3 months
  the time interval from the day of surgery to the day of chest tube removal
post-operative pulmonary function | 6, 12 and 24 months
  the pulmonary function at 6, 12, and 24 months post-operation

OTHER OUTCOMES:
pain score | 1, 3, and 7 days
  post-operative pain assessment during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Lee Jang-Ming, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ginsberg RJ, Rubinstein LV. Randomized trial of lobectomy versus limited resection for T1 N0 non-small cell lung cancer. Lung Cancer Study Group. Ann Thorac Surg. 1995 Sep;60(3):615-22; discussion 622-3. doi: 10.1016/0003-4975(95)00537-u. PMID 7677489
- [Result] Sienel W, Dango S, Kirschbaum A, Cucuruz B, Horth W, Stremmel C, Passlick B. Sublobar resections in stage IA non-small cell lung cancer: segmentectomies result in significantly better cancer-related survival than wedge resections. Eur J Cardiothorac Surg. 2008 Apr;33(4):728-34. doi: 10.1016/j.ejcts.2007.12.048. Epub 2008 Feb 7. PMID 18261918
- [Result] Kodama K, Doi O, Higashiyama M, Yokouchi H. Intentional limited resection for selected patients with T1 N0 M0 non-small-cell lung cancer: a single-institution study. J Thorac Cardiovasc Surg. 1997 Sep;114(3):347-53. doi: 10.1016/S0022-5223(97)70179-X. PMID 9305186
- [Result] Okada M, Yoshikawa K, Hatta T, Tsubota N. Is segmentectomy with lymph node assessment an alternative to lobectomy for non-small cell lung cancer of 2 cm or smaller? Ann Thorac Surg. 2001 Mar;71(3):956-60; discussion 961. doi: 10.1016/s0003-4975(00)02223-2. PMID 11269480